CLINICAL TRIAL: NCT00011609
Title: Clinical Evaluation of a Wheelchair Mounted Robotic Arm
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2311T
Record Dates: First submitted 2001-02-22; First posted 2001-02-26 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2001-01

CONDITIONS: Spinal Cord Injury
Keywords: Robotics; Activities of Daily Living; Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

INTERVENTIONS:
Device: Robotic Arm

SUMMARY:
The primary purpose of this project, is to evaluate the effect of a wheelchair mounted robotic arm (WMRA) to improve the functional independence of veterans with SCI.

The study will determine if the ability to perform marker tasks within the following four categories is improved after the 4 week training period using the robotic arm:

1. activities of daily living, 2. vocational tasks, 3. advanced tasks, and subject-specific tasks.

DETAILED DESCRIPTION:
The primary purpose of this project, is to evaluate the effect of a wheelchair mounted robotic arm (WMRA) to improve the functional independence of veterans with SCI.

The study will determine if the ability to perform marker tasks within the following four categories is improved after the 4 week training period using the robotic arm:

1. activities of daily living, 2. vocational tasks, 3. advanced tasks, and subject-specific tasks.

The secondary purposes of this project are the following: 1.Does quality of life (life satisfaction and health status) improve after a 4 week period of using the WMRA? 2. What are the perceived advantages of the WMRA to the veteran with SCI? Additionally, the study will evaluate the following: 1) ease of installation and usefulness of instructional manuals; 2) training requirements (time, tasks); 3) safety features; 4) reliability of the device; 5) home, community, and vocational applications; 6) user acceptability; 7) maintenance/ service; 8) portability; and possible modifications.

ELIGIBILITY:
Patients with spinal cord injuries

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2000-08; Study Completion 2001-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Fryer, Ph.D. Asst. Director — Department of Veterans Affairs, Program Analysis and Review Section (PARS), Rehabilitation Research & Development Service; Nancy Rocheleau, Program Analyst — Department of Veterans Affairs, Program Analysis and Review Section (PARS), Rehabilitation Research & Development Service
Locations (1):
- VAMC, Houston, Houston, Texas, United States